CLINICAL TRIAL: NCT07257939
Title: A Phase III Double-blind, Randomised, Placebo-controlled Study Investigating the Efficacy and Safety of NTI164 in Children and Young Adults With Autism Spectrum Disorder
Brief Title: NTI164 in Autism Spectrum Disorder
Acronym: HarmonyPlus
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fenix Innovation Group (Industry)
Collaborators: Neurotech International Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NTIASD3; FENASD3 (Other: Fenix Innovation Group)
Record Dates: First submitted 2025-11-17; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Autism; Autism Spectrum Disorder; Autism Disorder
Keywords: Cannabis; NTI164; Autism spectrum disorder
MeSH Terms: conditions — Autistic Disorder; Autism Spectrum Disorder; Marijuana Abuse

STUDY DESIGN:
Intervention Model Description: Double-blind, randomised, placebo-controlled, parallel
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All study team members will be blinded during the main treatment phase of this study (i.e up to Week 16). Only Clinical Trial Pharmacy staff will be unblinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active (Experimental): NTI164
  Interventions: Drug: NTI164
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NTI164 — A CBDA-dominant full-spectrum medicinal cannabis plant extract with extremely low THC.
  Other Names: FEN164
  Arms: Active
Drug: Placebo — Placebo oil suspension
  Arms: Placebo

SUMMARY:
This is a double-blind, randomised, placebo-controlled study investigating the efficacy of a full-spectrum medicinal cannabis plant extract on core and associated ASD symptoms over placebo. Participants will be randomly allocated to either NTI164 or placebo at a 1:1 ratio and blood samples will be collected and surveys completed at baseline and Week 16. This study will expand efficacy and safety data of NTI164 and provide additional mechanism of action data of NTI164 in this patient cohort.

DETAILED DESCRIPTION:
Participants will be recruited from Monash Health, Vic, Australia and will have a diagnosis of ASD Level II or III, as well as satisfying other inclusion/exclusion criteria. The primary objective is to assess efficacy of 16 weeks of daily oral administration of NTI164 on core ASD symptoms compared to placebo. The secondary objectives are to further expand the safety data of NTI164 in this patient cohort, and assess the changes in other associated symptoms of ASD following NTI164.

ELIGIBILITY:
Inclusion Criteria:

1. Participant is aged 6 years to 25 years (inclusive).
2. Participant is at a healthy weight at the discretion of the Principal Investigator.
3. Written informed consent from parent or legal guardian according to the local law.
4. Participants can comply with trial requirements.
5. According the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) criteria the participant has a diagnosis of Level II or III ASD confirmed by a validated assessment tool.
6. All treatments including medications and therapies for ASD related symptoms must have been stable for 12 weeks before enrolment and for the duration of the trial wherever possible.
7. Participants must be able to swallow liquid.
8. Consent giver must be able to understand the requirements of the study.

Exclusion Criteria:

1. Current diagnosis of bipolar disorder, psychosis, schizophrenia, schizoaffective disorder, or active major depression.
2. Has a diagnosis other than ASD that dominates the clinical presentation (e.g., ADHD).
3. Has a degenerative condition.
4. Changes in anticonvulsive therapy within the last 12 weeks.
5. Taking omeprazole, lansoprazole, tolbutamide, warfarin, sirolimus, everolimus, temsirolimus, tacrolimus, clobazam, repaglinide, pioglitazone, rosiglitazone, montelukast, bupropion, or efavirenz.
6. Currently using or has used recreational or medicinal cannabis, cannabinoid-based medications (including Sativex®, or Epidiolex®) within the 12 weeks prior to screening and is unwilling to abstain for the duration of the trial.
7. Participant has any known or suspected hypersensitivity to cannabinoids or any of the excipients.
8. Participant has moderately impaired hepatic function at screening, defined as serum alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 2 × upper limit of normal (ULN) or total bilirubin (TBL) > 2 × ULN. This criterion can only be confirmed once the laboratory results are available; participants enrolled into the trial who are later found to meet this criterion must be screen-failed.
9. Participant is male and fertile (i.e., after puberty unless permanently sterile by bilateral orchidectomy) unless willing to ensure that they use male contraception (condom) or remain sexually abstinent during the trial and for 12 weeks thereafter.
10. Participant is female and with childbearing potential (i.e., following menarche and until becoming postmenopausal for ≥ 12 consecutive months unless permanently sterile by hysterectomy, bilateral salpingectomy, or bilateral oophorectomy) unless willing to ensure that they use a highly effective method of birth control (e.g., hormonal contraception, intrauterine device/hormone-releasing system, bilateral tubal occlusion, vasectomised partner, sexual abstinence) during the trial and for 12 weeks thereafter.
11. Female participant who is pregnant (positive pregnancy test), lactating or planning pregnancy during the course of the trial or within 12 weeks thereafter.
12. Participant had brain surgery or traumatic brain injury within 1 year of screening.
13. Participant has any other significant disease or disorder which, in the opinion of the Investigator, may either put the participant, other participants, or site staff at risk because of participation in the trial, may influence the result of the trial, or may affect the participant's ability to take part in the trial.
14. Any abnormalities identified following a physical examination of the participant that, in the opinion of the Investigator, would jeopardise the safety of the participant if they took part in the trial.
15. Any history of suicidal behaviour (lifelong) or any suicidal ideation of type 4 or 5 on the Columbia-Suicide Severity Rating Scale (C-SSRS) in the last 12 weeks or at screening or randomisation.
16. Participant has donated blood during the past 12 weeks and is unwilling to abstain from donation of blood during the trial.
17. Participant has any known or suspected history of alcohol or substance abuse or positive drugs of abuse test at screening (not justified by a known concurrent medication).
18. Participant has previously been enrolled into this trial.
19. Participant has plans to travel outside their country of residence during the trial, unless the participant has confirmation that the product is permitted in the destination country/state.

Ages: 6 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 98 (Estimated)
Dates: Start 2026-07-01 (Estimated); Primary Completion 2029-07-01 (Estimated); Study Completion 2030-07-01 (Estimated)

PRIMARY OUTCOMES:
Social Responsiveness Scale, 2nd Edition (SRS-2) | Baseline, Week 16
  Captures overall change in core ASD symptoms across domains including social awareness, social cognition, social communication, social motivation, and restricted and repetitive behaviours. Scores are between 0-195, and higher scores indicate greater impairment.

SECONDARY OUTCOMES:
Vineland Adaptive Behaviour Scales, 3rd Edition (Vineland-3) | Baseline, Week 16
  Used to measure functioning across 3 core domains, Communication, Daily Living Skills, and Socialisation, as well as 2 optional domains, Motor Skills and Maladaptive Behaviour. The core domains sum to a total Adaptive Behaviour Composite. Scores are between 20-160, higher scores indicate better outcomes.
Clinical Global Impression - Improvement (CGI-I) | Baseline, Week 16
  Provides a clinician-rated global assessment of improvement at a given time point following an intervention. 1-3 = improvement, 4 = no change, 5-7 = worsening.
Clinical Global Impression - Severity (CGI-S) | Baseline, Week 16
  Evaluates a clinician's impression of disease severity at a given time point from a scale of 1-7. A higher score indicates greater impairment/disease severity.
Anxiety, Depression, and Mood Scale (ADAMS) | Baseline, Week 16
  Measures emotional and behavioural disturbances frequently comorbid with ASD. Assesses 5 domains (Manic/hyperactive Behaviour, Depressed Mood, Social Avoidance, General Anxiety, and Compulsive Behaviour). Scores are between 0-84, with higher scores indicating greater impairment.
Autism Family Experience Questionnaire (AFEQ) | Baseline, Week 16
  Captures caregiver perceptions of changes in family impact, child wellbeing, and support burden. Scores range from 48-240, with higher scores indicating worse family outcomes.
Sleep Disturbances Scale for Children (SDSC) | Baseline, Week 16
  Evaluates treatment-related changes in sleep quality and sleep-wake behaviours. Assesses 6 domains (Disorders of Initiating and Maintaining Sleep, Sleep Breathing Disorders, Disorders of Arousal, Sleep Wake Transition Disorders, Disorders of Excessive Somnolence, and Sleep Hyperhidrosis). Scores range from 26-130, with higher scores indicating greater impairment and issues around sleep.
EQ-5D-Y-5L | Baseline, Week 16
  Measures broader wellbeing and day-to-day function, as well as quality of life (QoL), from a caregiver-reported perspective. Assesses health in 5 domains (Mobility, Usual Activities, Self-care, Pain/discomfort, and Anxiety/depression), and QoL. Scores range from 0-1, with 0 = the worst health possible and 1 = the best possible health state. The higher the score, the better the health state.
Anxiety Scale for Children with ASD, Parent edition (ASC-ASD-P) | Baseline, Week 16
  Evaluates changes in anxiety symptoms and emotional regulation. It is used to detect symptoms of anxiety in youth with ASD and assesses 4 domains (Performance Anxiety, Uncertainty, Anxious Arousal, and Separation Anxiety). Scores range from 0-72, with higher scores indicating greater impairment.
Aberrant Behaviour Checklist (ABC) | Baseline, Week 16
  Assesses challenging behaviours and behavioural regulation relevant to ASD functioning. Measures impairment across 5 domains (Irritability, Lethargy/social Withdrawal, Stereotypic Behaviour, Hyperactivity/non-compliance, and Inappropriate Speech. Scores range from 0-174, with higher scores indicating greater impairment.

OTHER OUTCOMES:
Research samples - transcriptomics | Baseline, Week 16
  To further clarify the mechanism of action of NTI164, both bulk and single-cell RNA sequencing will be performed on peripheral blood mononuclear cells (PBMCs) from patients at specified time points. This will provide additional information regarding which genes are being expressed in patients at either abnormally low or high levels compared to a non-ASD population, and the effects NTI164 has on gene expression. This workflow includes RNA extraction, depletion of ribosomal RNA via hybrid capture, library preparation, and sequencing. Cleaned sequence reads will then be aligned against the Homo sapiens genome (Build version hg38) and STAR aligner (v2.5.3a) will be used to map unique reads to the genomic sequences. This is exploratory so genes of interest cannot be identified in advance.
Research bloods - proteomics (and phosphoproteomics) | Baseline, Week 16
  To further clarify the mechanism of action of NTI164, proteomics and phosphoproteomics will be performed on peripheral blood mononuclear cells (PBMCs) from patients at specified time points. This will provide additional information regarding which proteins are being expressed at either abnormally low or high levels compared to a non-ASD population, as well as how extensively these proteins are phosphorylated compared to a non-ASD population, and the effects NTI164 has on protein expression and phosphorylation. Samples will be tagged using the TMTpro system and hydrophilic ion liquid chromatography fractionation performed. This is exploratory so proteins of interest cannot be identified in advance.
Research bloods - Methylomics | Baseline, Week 16
  To further clarify the mechanism of action of NTI164, methylomics will be performed on whole blood from patients at specified time points. This will provide additional information on methylation patterns (e.g. addition of a methyl group to histones or DNA) in patients compared to non-patients, and how NTI164 effects this type of epigenetic modification and how genes of interest may be regulated. This is exploratory so patterns of interest cannot be identified in advance. Genome-wide methylation will be assessed using the Illumina MethylationEPIC v2.0 BeadChip (or the latest version if a new version is available to the study team at the time of analysis).
Research bloods - cytokine assay | Baseline, Week 16
  To further clarify the mechanism of action of NTI164, a cytokine assay investigating a panel of inflammatory markers will be performed on plasma from patients at specified time points. The cytokine assay will likely be the LEGENDplex Human Neuroinflammation Panel 1 (13 plex). Cytokines investigated with this panel include VILIP-1, CCL2, sTREM-2, b-NGF, TGF-b1, TNF-a, IL-6, s-TREM-1, sRAGE, CX3CL1, VEGF, BDNF, and IL-18.

CONTACTS AND LOCATIONS:
Locations (1):
- Monash Health, Clayton, Victoria, Australia